CLINICAL TRIAL: NCT03384121
Title: Rifampin to Reduce Elevated Levels of Blood and Urine Calcium in Patients With Idiopathic Infantile Hypercalcemia
Brief Title: The Antibiotic Rifampin to Reduce High Levels of Blood and Urine Calcium in IIH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital of Philadelphia (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Cures Within Reach (Other)
Responsible Party: Principal Investigator, Etienne Sochett, Staff Endocrinologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000057141
Record Dates: First submitted 2017-12-13; First posted 2017-12-27 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Idiopathic Infantile Hypercalcemia - Mild Form
Keywords: CYP24A1; Nephrocalcinosis; Hypercalcemia; Hypercalcuria
MeSH Terms: conditions — Nephrocalcinosis; Hypercalcemia; Hypercalciuria | interventions — Rifampin; Suspensions

STUDY DESIGN:
Intervention Model Description: This is a phase 1 pilot study whereby all participants start the study at a starting dose 5mg/kg/day (at study visit 2) for two months, and those that do not respond to 5mg/kg/day, otherwise known as non-responders, will receive a higher dose of 10 mg/kg/day (at study visit 4) for another two months. Recruited patients will be followed prospectively for a total of 6-11 months. This will include 2 months of observation, 2 months of receiving the starting dose of rifampin of 5mg/kg/day with a maximum dose of 600mg/day followed by a 2 month washout phase. The efficacy of the starting dose of rifampin will be determined prior to proceeding only in non-responders to the higher dose of 10 mg/kg/day with a maximum dose of 600 mg/day.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rifampin (Experimental): All subjects
  Interventions: Drug: Rifampin 150 mg, 300 mg capsules and 25 mg/mL oral suspension

INTERVENTIONS:
Drug: Rifampin 150 mg, 300 mg capsules and 25 mg/mL oral suspension — Starting Dose (V2): 5 mg/kg/day (max 600mg/day) orally for 2 months followed by a 2 month washout period V4: After washout period, only Non-responders will escalate dose to 10 mg/kg/day (max 600mg/day) orally for 2 months
  Other Names: Rifadin, Rofact, Rifampicin

SUMMARY:
Idiopathic infantile hypercalcemia(IIH) is a rare,genetic disorder of mineral metabolism. Biallelic loss of functions mutations of CYP24A1, the gene encoding the 24-hydroxylase enzyme that represents the principal pathway for inactivation of vitamin D metabolites, cause the most common and severe form of IIH.Investigators have preliminary data supporting a novel therapeutic approach to suggest rifampin as an investigational drug to induce over-expression of CYP3A4, an important enzyme that provides an alternate catabolic pathway for inactivation of vitamin D metabolites. In this study, investigators will recruit 5 patients with biallelic inactivating mutations of CYP24A1. Participants will be followed prospectively for a total 6-11 months. This will include 2 months of observation, 2 months of receiving the starting dose of rifampin, followed by 2 month washout phase. Efficacy of the starting dose of rifampin will be determined prior to proceeding only in non responders to the escalation dose of rifampin 10mg/kg/day.

DETAILED DESCRIPTION:
Idiopathic infantile hypercalcemia(IIH) is a rare,genetic disorder of mineral metabolism characterized by severe hypercalcemia and/or hypercalciuria, suppressed serum levels of parathyroid hormone (PTH), elevated levels of the active vitamin D metabolite, 1,25(OH)2D, and nephrocalcinosis. Biallelic loss of functions mutations of CYP24A1, the gene encoding the 24-hydroxylase enzyme that represents the principal pathway for inactivation of vitamin D metabolites, cause the most common and severe form of IIH.

Investigators have preliminary data supporting a novel therapeutic approach to suggest rifampin as an investigational drug to induce over-expression of CYP3A4, an important P450 microsomal enzyme that is expressed in the liver and intestine. When CYP3A4 is induced, the increased enzyme activity provides an alternative catabolic pathway for inactivation of vitamin D metabolites. The purpose of this study is to obtain results and support for an open label, escalating dose study to assess the effect, safety, and tolerability of once daily oral rifampin for two months in participants with IIH due to inactivating mutations in CYP24A1.

In this study, Investigators will recruit 5 patients with biallelic inactivating mutations of CYP24A1. Participants will be followed prospectively for a total 6-11 months. This will include 2 months of observation, 2 months of receiving the starting dose of rifampin, followed by 2 month washout phase. Efficacy of the starting dose of rifampin will be determined prior to proceeding only in non responders to the escalation dose of rifampin 10mg/kg/day. In addition to determining if this treatment is efficacious in reducing elevated serum and urinary calcium in patients, it will be determined if there is a dose effect of rifampin. As well, detailed measurements of vitamin D metabolites will determine if rifampin reduces hypercalcemia through increased CYP3A4 activity.

ELIGIBILITY:
Inclusion Criteria:

* all patients between 6 months- 17 years of age with the clinical phenotype of idiopathic infantile hypercalcemia
* Biochemical evidence of this disorder: Serum calcium>upper limit of the reference age for range; high, 1,25 (OH)D; reduced PTH, reduced 24,25(OH)2D, and suppresses 24,1,25 (OH)2D, normal serum creatinine, AST, and ALT with or without
* biallelic inactivating mutations of CYP24A1
* mutations in newly published genes which are shown during the course of the study to cause an inappropriate increase in 1,25 (OH)2D

Exclusion Criteria:

* Allergy to rifampin or related medications
* Pregnancy or breastfeeding
* Significant cardiac, hepatic, or endocrine comorbidities
* Taking any medications/foods known to interact with CYP3A4 or 1,25 (OH)D
* Parents or guardians or subjects who in the opinion of the Investigator may be non compliant with study schedules or procedures
* Other comorbidities considered unsuitable by the investigator, including TB

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Serum Calcium | 40 weeks
  Measured at baseline and every 2 months (8 weeks)
Change in Serum Parathyroid Hormone | 40 weeks
  measured at baseline and every 2 months ( 8 weeks)
Change in Urinary calcium excretion | 40 weeks
  Measured at baseline and every 2 months( 8 weeks)

SECONDARY OUTCOMES:
Nephrocalcinosis | 40 weeks
  Renal ultrasound performed before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Sochett, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] LIGHTWOOD R, STAPLETON T. Idiopathic hypercalcaemia in infants. Lancet. 1953 Aug 1;265(6779):255-6. doi: 10.1016/s0140-6736(53)90187-1. No abstract available. PMID 13070618
- [Background] CREERY RD, NEILL DW. Idiopathic hypercalcaemia in infants with failure to thrive. Lancet. 1954 Jul 17;267(6829):110-4. doi: 10.1016/s0140-6736(54)90094-x. No abstract available. PMID 13175473
- [Background] Masuda S, Byford V, Arabian A, Sakai Y, Demay MB, St-Arnaud R, Jones G. Altered pharmacokinetics of 1alpha,25-dihydroxyvitamin D3 and 25-hydroxyvitamin D3 in the blood and tissues of the 25-hydroxyvitamin D-24-hydroxylase (Cyp24a1) null mouse. Endocrinology. 2005 Feb;146(2):825-34. doi: 10.1210/en.2004-1116. Epub 2004 Oct 21. PMID 15498883
- [Background] Schlingmann KP, Kaufmann M, Weber S, Irwin A, Goos C, John U, Misselwitz J, Klaus G, Kuwertz-Broking E, Fehrenbach H, Wingen AM, Guran T, Hoenderop JG, Bindels RJ, Prosser DE, Jones G, Konrad M. Mutations in CYP24A1 and idiopathic infantile hypercalcemia. N Engl J Med. 2011 Aug 4;365(5):410-21. doi: 10.1056/NEJMoa1103864. Epub 2011 Jun 15. PMID 21675912
- [Background] Dauber A, Nguyen TT, Sochett E, Cole DE, Horst R, Abrams SA, Carpenter TO, Hirschhorn JN. Genetic defect in CYP24A1, the vitamin D 24-hydroxylase gene, in a patient with severe infantile hypercalcemia. J Clin Endocrinol Metab. 2012 Feb;97(2):E268-74. doi: 10.1210/jc.2011-1972. Epub 2011 Nov 23. PMID 22112808
- [Background] KENNY FM, ACETO T Jr, PURISCH M, HARRISON HE, HARRISON HC, BLIZZARD RM. Metabolic studies in a patient with idiopathic hypercalcemia of infancy. J Pediatr. 1963 Apr;62:531-7. doi: 10.1016/s0022-3476(63)80010-4. No abstract available. PMID 14031980
- [Background] Pronicka E, Kulczycka H, Rowinska E, Konopinska A, Kansy J, Lorenc R. [Idiopathic hypercalcemia as a syndrome of hypersensitivity to vitamin D3 in 19 infants]. Pediatr Pol. 1985 Apr;60(4):288-94. No abstract available. Polish. PMID 2995910
- [Background] SMITH DW, BLIZZARD RM, HARRISON HE. Idiopathic hypercalcemia; a case report with assays of vitamin D in the serum. Pediatrics. 1959 Aug;24(2):258-69. No abstract available. PMID 13674824
- [Background] Wolf P, Muller-Sacherer T, Baumgartner-Parzer S, Winhofer Y, Kroo J, Gessl A, Luger A, Krebs M. A Case of "Late-Onset" Idiopathic Infantile Hypercalcemia Secondary to Mutations in the CYP24A1 Gene. Endocr Pract. 2014 May;20(5):e91-5. doi: 10.4158/EP13479.CR. PMID 24518185
- [Background] Tray KA, Laut J, Saidi A. Idiopathic Infantile Hypercalcemia, Presenting in Adulthood--No Longer Idiopathic Nor Infantile: Two Case Reports and Review. Conn Med. 2015 Nov-Dec;79(10):593-7. PMID 26731879
- [Background] Nesterova G, Malicdan MC, Yasuda K, Sakaki T, Vilboux T, Ciccone C, Horst R, Huang Y, Golas G, Introne W, Huizing M, Adams D, Boerkoel CF, Collins MT, Gahl WA. 1,25-(OH)2D-24 Hydroxylase (CYP24A1) Deficiency as a Cause of Nephrolithiasis. Clin J Am Soc Nephrol. 2013 Apr;8(4):649-57. doi: 10.2215/CJN.05360512. Epub 2013 Jan 4. PMID 23293122
- [Background] Cools M, Goemaere S, Baetens D, Raes A, Desloovere A, Kaufman JM, De Schepper J, Jans I, Vanderschueren D, Billen J, De Baere E, Fiers T, Bouillon R. Calcium and bone homeostasis in heterozygous carriers of CYP24A1 mutations: A cross-sectional study. Bone. 2015 Dec;81:89-96. doi: 10.1016/j.bone.2015.06.018. Epub 2015 Jun 25. PMID 26117226
- [Background] Prosser DE, Jones G. Enzymes involved in the activation and inactivation of vitamin D. Trends Biochem Sci. 2004 Dec;29(12):664-73. doi: 10.1016/j.tibs.2004.10.005. PMID 15544953
- [Background] Cheng JB, Levine MA, Bell NH, Mangelsdorf DJ, Russell DW. Genetic evidence that the human CYP2R1 enzyme is a key vitamin D 25-hydroxylase. Proc Natl Acad Sci U S A. 2004 May 18;101(20):7711-5. doi: 10.1073/pnas.0402490101. Epub 2004 May 5. PMID 15128933
- [Background] Bergwitz C, Juppner H. Regulation of phosphate homeostasis by PTH, vitamin D, and FGF23. Annu Rev Med. 2010;61:91-104. doi: 10.1146/annurev.med.051308.111339. PMID 20059333
- [Background] Shimada T, Hasegawa H, Yamazaki Y, Muto T, Hino R, Takeuchi Y, Fujita T, Nakahara K, Fukumoto S, Yamashita T. FGF-23 is a potent regulator of vitamin D metabolism and phosphate homeostasis. J Bone Miner Res. 2004 Mar;19(3):429-35. doi: 10.1359/JBMR.0301264. Epub 2003 Dec 29. PMID 15040831
- [Background] Levine MA. Normal mineral homeostasis. Interplay of parathyroid hormone and vitamin D. Endocr Dev. 2003;6:14-33. doi: 10.1159/000072764. No abstract available. PMID 12964423
- [Background] Christakos S, Dhawan P, Verstuyf A, Verlinden L, Carmeliet G. Vitamin D: Metabolism, Molecular Mechanism of Action, and Pleiotropic Effects. Physiol Rev. 2016 Jan;96(1):365-408. doi: 10.1152/physrev.00014.2015. PMID 26681795
- [Background] Dusso AS, Gomez-Alonso C, Cannata-Andia JB. The hypercalcaemia of CYP24A1 inactivation: new ways to improve diagnosis and treatment. Clin Kidney J. 2015 Aug;8(4):456-8. doi: 10.1093/ckj/sfv058. Epub 2015 Jul 6. PMID 26251717
- [Background] Curtis KM, Aenlle KK, Roos BA, Howard GA. 24R,25-dihydroxyvitamin D3 promotes the osteoblastic differentiation of human mesenchymal stem cells. Mol Endocrinol. 2014 May;28(5):644-58. doi: 10.1210/me.2013-1241. Epub 2014 Mar 5. PMID 24597546
- [Background] Greising DM, Schwartz Z, Posner GH, Sylvia VL, Dean DD, Boyan BD. A-ring analogues of 1, 25-(OH)2D3 with low affinity for the vitamin D receptor modulate chondrocytes via membrane effects that are dependent on cell maturation. J Cell Physiol. 1997 Jun;171(3):357-67. doi: 10.1002/(SICI)1097-4652(199706)171:33.0.CO;2-7. PMID 9180905
- [Background] Nguyen M, Boutignon H, Mallet E, Linglart A, Guillozo H, Jehan F, Garabedian M. Infantile hypercalcemia and hypercalciuria: new insights into a vitamin D-dependent mechanism and response to ketoconazole treatment. J Pediatr. 2010 Aug;157(2):296-302. doi: 10.1016/j.jpeds.2010.02.025. Epub 2010 Apr 14. PMID 20394945
- [Background] Sayers J, Hynes AM, Srivastava S, Dowen F, Quinton R, Datta HK, Sayer JA. Successful treatment of hypercalcaemia associated with a CYP24A1 mutation with fluconazole. Clin Kidney J. 2015 Aug;8(4):453-5. doi: 10.1093/ckj/sfv028. Epub 2015 May 25. PMID 26251716
- [Background] Wang Z, Lin YS, Zheng XE, Senn T, Hashizume T, Scian M, Dickmann LJ, Nelson SD, Baillie TA, Hebert MF, Blough D, Davis CL, Thummel KE. An inducible cytochrome P450 3A4-dependent vitamin D catabolic pathway. Mol Pharmacol. 2012 Apr;81(4):498-509. doi: 10.1124/mol.111.076356. Epub 2011 Dec 28. PMID 22205755
- [Background] Xu Y, Hashizume T, Shuhart MC, Davis CL, Nelson WL, Sakaki T, Kalhorn TF, Watkins PB, Schuetz EG, Thummel KE. Intestinal and hepatic CYP3A4 catalyze hydroxylation of 1alpha,25-dihydroxyvitamin D(3): implications for drug-induced osteomalacia. Mol Pharmacol. 2006 Jan;69(1):56-65. doi: 10.1124/mol.105.017392. Epub 2005 Oct 5. PMID 16207822
- [Background] Wang Z, Wong T, Hashizume T, Dickmann LZ, Scian M, Koszewski NJ, Goff JP, Horst RL, Chaudhry AS, Schuetz EG, Thummel KE. Human UGT1A4 and UGT1A3 conjugate 25-hydroxyvitamin D3: metabolite structure, kinetics, inducibility, and interindividual variability. Endocrinology. 2014 Jun;155(6):2052-63. doi: 10.1210/en.2013-2013. Epub 2014 Mar 18. PMID 24641623
- [Background] Wang Z, Lin YS, Dickmann LJ, Poulton EJ, Eaton DL, Lampe JW, Shen DD, Davis CL, Shuhart MC, Thummel KE. Enhancement of hepatic 4-hydroxylation of 25-hydroxyvitamin D3 through CYP3A4 induction in vitro and in vivo: implications for drug-induced osteomalacia. J Bone Miner Res. 2013 May;28(5):1101-16. doi: 10.1002/jbmr.1839. PMID 23212742
- [Background] Kreis B, Pretet S, Birenbaum J, Guibout P, Hazeman JJ, Orin E, Perdrizet S, Weil J. Two three-month treatment regimens for pulmonary tuberculosis. Bull Int Union Tuberc. 1976;51(1):71-5. No abstract available. PMID 1030315
- [Background] Long MW, Snider DE Jr, Farer LS. U.S. Public Health Service Cooperative trial of three rifampin-isoniazid regimens in treatment of pulmonary tuberculosis. Am Rev Respir Dis. 1979 Jun;119(6):879-94. doi: 10.1164/arrd.1979.119.6.879. PMID 110184
- [Background] Poole G, Stradling P, Worlledge S. Potentially serious side effects of high-dose twice-weekly rifampicin. Br Med J. 1971 Aug 7;3(5770):343-7. doi: 10.1136/bmj.3.5770.343. PMID 5314737
- [Background] Boeree MJ, Diacon AH, Dawson R, Narunsky K, du Bois J, Venter A, Phillips PP, Gillespie SH, McHugh TD, Hoelscher M, Heinrich N, Rehal S, van Soolingen D, van Ingen J, Magis-Escurra C, Burger D, Plemper van Balen G, Aarnoutse RE; PanACEA Consortium. A dose-ranging trial to optimize the dose of rifampin in the treatment of tuberculosis. Am J Respir Crit Care Med. 2015 May 1;191(9):1058-65. doi: 10.1164/rccm.201407-1264OC. PMID 25654354
- [Background] Thacher TD, Fischer PR, Singh RJ, Roizen J, Levine MA. CYP2R1 Mutations Impair Generation of 25-hydroxyvitamin D and Cause an Atypical Form of Vitamin D Deficiency. J Clin Endocrinol Metab. 2015 Jul;100(7):E1005-13. doi: 10.1210/jc.2015-1746. Epub 2015 May 5. PMID 25942481
- [Background] Wang Z, Senn T, Kalhorn T, Zheng XE, Zheng S, Davis CL, Hebert MF, Lin YS, Thummel KE. Simultaneous measurement of plasma vitamin D(3) metabolites, including 4beta,25-dihydroxyvitamin D(3), using liquid chromatography-tandem mass spectrometry. Anal Biochem. 2011 Nov 1;418(1):126-33. doi: 10.1016/j.ab.2011.06.043. Epub 2011 Jul 13. PMID 21784054
- [Background] O'Brien RJ, Long MW, Cross FS, Lyle MA, Snider DE Jr. Hepatotoxicity from isoniazid and rifampin among children treated for tuberculosis. Pediatrics. 1983 Oct;72(4):491-9. PMID 6604257
- [Background] Saukkonen JJ, Cohn DL, Jasmer RM, Schenker S, Jereb JA, Nolan CM, Peloquin CA, Gordin FM, Nunes D, Strader DB, Bernardo J, Venkataramanan R, Sterling TR; ATS (American Thoracic Society) Hepatotoxicity of Antituberculosis Therapy Subcommittee. An official ATS statement: hepatotoxicity of antituberculosis therapy. Am J Respir Crit Care Med. 2006 Oct 15;174(8):935-52. doi: 10.1164/rccm.200510-1666ST. PMID 17021358